CLINICAL TRIAL: NCT05764473
Title: Dietary Patterns, Cardiometabolic Risk Factors and Menopause Symptoms in a Sample of UK Women - A Randomised Cross-over Parallel Trial
Brief Title: Diet, Cardiometabolic Risk (CM) and Menopause Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chester (Other)
Responsible Party: Principal Investigator, Tanja Harrison, Lecturer in Public Health Nutrition, University of Chester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MenoUoC
Record Dates: First submitted 2023-02-13; First posted 2023-03-10 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Syndrome, Protection Against; Menopause
Keywords: menopause; peri-menopause; post-menopause; vasomotor symptoms; cardiometabolic risk; Mediterranean Diet; MedDiet; Ultimate Cholesterol Lowering Plan; UCLP; Portfolio diet; diet quality
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: 12-week randomised cross-over parallel trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Med/UCLP) (Experimental): Following the Mediterranean Diet for six weeks, then following the Ultimate Cholesterol Lowering Plan for six weeks.
  Food diaries collected at baseline, week 2, week 4, week 6, week 8, week 10, week 12.
  Cardiometabolic risk markers, menopause symptoms and physical activity collected at baseline, week 6, week 12.
  Interventions: Other: The impact of MedDiet on cardiometabolic risk factors and menopause symptoms; Other: The impact of UCLP on cardiometabolic risk factors and menopause symptoms
- B (ULCP/Med) (Experimental): Following the Ultimate Cholesterol Lowering Plan for six weeks, then following the Mediterranean Diet for six weeks.
  Food diaries collected at baseline, week 2, week 4, week 6, week 8, week 10, week 12.
  Cardiometabolic risk markers, menopause symptoms and physical activity collected at baseline, week 6, week 12.
  Interventions: Other: The impact of MedDiet on cardiometabolic risk factors and menopause symptoms; Other: The impact of UCLP on cardiometabolic risk factors and menopause symptoms

INTERVENTIONS:
Other: The impact of MedDiet on cardiometabolic risk factors and menopause symptoms — 12-week randomised parallel cross-over study with 32 participants. Impact of diet on CMR factors and menopause symptoms will be explored with diet quality and adherence to diet determined via diet quality indices for MedDiet and Portfolio diet.
Other: The impact of UCLP on cardiometabolic risk factors and menopause symptoms — 12-week randomised parallel cross-over study with 32 participants. Impact of diet on CMR factors and menopause symptoms will be explored with diet quality and adherence to diet determined via diet quality indices for MedDiet and Portfolio diet.

SUMMARY:
This research will explore the question 'What impact do the Mediterranean Diet (MedDiet) and the Heart UK Ultimate Cholesterol Lowering Plan (UCLP) Menopause have on cardiometabolic risk factors and the frequency and severity of menopause symptoms? This is a randomised cross-over parallel trial of 12 weeks duration. Participants are women undergoing or having completed the menopause transition.

DETAILED DESCRIPTION:
Group 1 will first follow the MedDiet pattern for six weeks and then follow the UCLP diet pattern for six weeks. Group 2 will also follow both diet patterns but in the opposite order.

Week 0 will be the baseline, week 6 will be the interim point and week 12 will be the endpoint.

Data collection Some data will be collected at the University of Chester laboratories, including anthropometric measurements, blood pressure and blood samples. A small fasted blood sample will be collected via finger prick (Alere Cholestech LDX® Analyzer (Alere San Diego Inc. USA)). Participants will also be talked through the guidance notes for the diets at this point. Other data, food diaries and a questionnaire asking about recent physical activity and menopause symptoms will be completed online.

Demographics At baseline participants will be asked to complete a brief questionnaire to answer a few demographic questions, including date of birth, ethnicity, income category, level of education, whether (and if so which) using any form of hormone replacement therapy (HRT) or contraception. Participants will be asked at interim and endpoint whether there have been any recent changes with regards to HRT and contraception methods.

Dietary intake Participants will be asked to complete a total of seven four-day food diaries. The first diary will be completed in the week before participants attend their first appointment in the laboratory. This diary will give a snapshot of the participants' habitual diet prior to joining the intervention. The other four-day food diaries will be completed in weeks 2, 4, 6, 8, 10 and 12.

Physical activity Data on physical activity over the previous four-week period will be collected at baseline, interim point and endpoint. Participants will be asked to complete the Recent Physical Activity Questionnaire (RPAQ).

Data analysis Blood sample Blood samples will be used to assess whether participants have

* elevated total cholesterol levels (>5 mmol/L)
* elevated LDL cholesterol levels (>3.0 mmol/L)
* elevated non-HDL cholesterol levels (>4 mmol/L)
* decreased HDL cholesterol levels (<1.3 mmol/L)
* elevated triglyceride levels (>1.7 mmol/L)
* elevated glucose levels (> 5.6 mmol/L)

HDL-C, glucose and triglyceride levels will also be used together with waist circumference and blood pressure data to assess whether participants present with metabolic syndrome at baseline, interim point and endpoint according to the definition of Alberti et al. (2009)

Dietary intake Food diary data will be analysed using the dietary assessment software Nutritics (2021).

The data from the analysis will also be used to identify the intake of phytoestrogen-rich foods (associated with milder menopause symptoms) and the average intake of phytoestrogens.

Dietary adherence and diet quality Following on from the analysis of the food diaries adherence to the MedDiet will be assessed by applying the Mediterranean Diet Score.

Adherence to the UCLP Menopause will be assessed by applying an amended version of the Portfolio Diet Score. The scoring system will be slightly adjusted where there are differences in terms of amounts to be consumed of the four portfolio foods.

Physical activity Each activity across the four domains of the RPAQ has a MET score assigned based on Ainsworth et al.'s (2011) updated Compendium of Physical Activities to categorise the activity as sedentary, light, moderate or vigorous intensity. Recoding of the completed RPAQ will follow the script devised by Medical Research Council (MRC) Epidemiology Unit (Scott et al., 2013; available to download at www.mrc-epid.cam.ac.uk/physical-activity-downloads/).

Statistical analysis Descriptive statistics (means (M) and standard deviation (SD)) will be produced for all data collected. Data will also be analysed for correlations between dietary intake, diet quality and changes to cardiometabolic risk (CMR) and to menopause symptoms. Mixed ANOVAs and linear and logistic regression analysis will also be employed. If necessary data will be adjusted for factors, such as physical activity, ethnicity, HRT intake, contraceptive intake, educational level and income category.

ELIGIBILITY:
Inclusion Criteria:

* over the past year presented with any of the following

  1. Irregular periods or no periods at all
  2. Night sweats
  3. Hot flushes
  4. Sleeplessness
  5. Brain fog
  6. Increased anxiety
  7. Joint pain
  8. Changes to hair or skin

     Exclusion Criteria:
* Ever had an eating disorder
* Ever diagnosed with cardiovascular disease or type 2 diabetes
* Ever diagnosed with kidney disease
* Current smoker
* Triglyceride levels of ≥ 5.7 mmol/L at baseline
* Glucose levels of ≥ 7 mmol/L at baseline
* Diastolic blood pressure of ≥ 100 mmHg at baseline
* Systolic blood pressure of ≥ 160 mmHg at baseline

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change Total cholesterol baseline-interim point | 6 weeks
  Change from baseline total cholesterol concentrations at 6 weeks
Change Total cholesterol baseline-endpoint | 12 weeks
  Change from baseline total cholesterol concentrations at 12 weeks
Change Total cholesterol interim point - endpoint | 6 weeks
  Change from interim point total cholesterol concentrations at 12 weeks
Change HDL cholesterol baseline - interim point | 6 weeks
  Change from baseline HDL cholesterol concentrations at 6 weeks
Change HDL cholesterol baseline - endpoint | 12 weeks
  Change from baseline HDL cholesterol concentrations at 12 weeks
Change HDL cholesterol interim point - endpoint | 6 weeks
  Change from interim point HDL cholesterol concentrations at 12 weeks
Change LDL cholesterol baseline-interim point | 6 weeks
  Change from baseline LDL cholesterol concentrations at 6 weeks
Change LDL cholesterol baseline - endpoint | 12 weeks
  Change from baseline LDL cholesterol concentrations at 12 weeks
Change LDL cholesterol interim point - endpoint | 6 weeks
  Change from interim point LDL cholesterol concentrations at 12 weeks
Change non-HDL cholesterol baseline - interim point | 6 weeks
  Change from baseline non-HDL cholesterol concentrations at 6 weeks
Change non-HDL cholesterol baseline - endpoint | 12 weeks
  Change from baseline non-HDL cholesterol concentrations at 12 weeks
Change non-HDL cholesterol interim point - endpoint | 6 weeks
  Change from interim point non-HDL cholesterol concentrations at 12 weeks
Change triglycerides baseline - interim point | 6 weeks
  Change from baseline triglyceride concentrations at 6 weeks
Change triglycerides - baseline - endpoint | 12 weeks
  Change from baseline triglyceride concentrations at 12 weeks
Change triglycerides interim point - endpoint | 6 weeks
  Change from interim point triglyceride concentrations at 12 weeks
Change blood glucose baseline - interim point | 6 weeks
  Change from baseline blood glucose concentrations at 6 weeks
Change blood glucose baseline - endpoint | 12 weeks
  Change from baseline blood glucose concentrations at 12 weeks
Change blood glucose interim point - endpoint | 6 weeks
  Change from interim point blood glucose concentrations at 12 weeks
Change Systolic and diastolic blood pressure baseline - interim point | 6 weeks
  Change from baseline systolic and diastolic blood pressure at 6 weeks
Change Systolic and diastolic blood pressure baseline - endpoint | 12 weeks
  Change from baseline blood glucose concentrations at 12 weeks
Change Systolic and diastolic blood pressure - interim point - endpoint | 6 weeks
  Change from interim point blood glucose concentrations at 12 weeks
Change Body mass index - baseline - interim point | 6 weeks
  Change from baseline body mass index at 6 weeks
Change Body mass index baseline - endpoint | 12 weeks
  Change from baseline body mass index at 12 weeks
Change Body mass index - interim point - endpoint | 6 weeks
  Change from interim point body mass index at 12 weeks
Change Waist circumference baseline - interim point | 6 weeks
  Change from baseline waist circumference at 6 weeks
Change Waist circumference baseline - endpoint | 12 weeks
  Change from baseline waist circumference at 12 weeks
Change Waist circumference interim point - endpoint | 6 weeks
  Change from interim point waist circumference at 12 weeks
Change Waist-hip ratio baseline - interim point | 6 weeks
  Change from baseline waist-hip ratio at 6 weeks
Change Waist-hip ratio baseline - endpoint | 12 weeks
  Change from baseline waist-hip ratio at 12 weeks
Change Waist-hip ratio interim point - endpoint | 6 weeks
  Change from interim point waist-hip ratio at 12 weeks
Change Waist-height ratio baseline - interim point | 6 weeks
  Change from baseline waist-height ratio at 6 weeks
Change Waist-height ratio baseline - endpoint | 12 weeks
  Change from baseline waist-height ratio at 12 weeks
Change Waist-height ratio interim point - endpoint | 6 weeks
  Change from interim point waist-height ratio at 12 weeks

SECONDARY OUTCOMES:
Change Frequency of menopause symptoms baseline - interim point | 6 weeks
  Change from baseline frequency of menopause symptoms at 6 weeks on a scale from 0 to 21 on the Greene Climacteric Scale. Higher Scores indicate higher frequency.
Change Frequency of menopause symptoms baseline - endpoint | 12 weeks
  Change from baseline frequency of menopause symptoms at 12 weeks on a scale from 0 to 21 on the Greene Climacteric Scale. Higher Scores indicate higher frequency.
Change Frequency of menopause symptoms - interim point - endpoint | 6 weeks
  Change from interim point frequency of menopause symptoms at 12 weeks on a scale from 0 to 21 on the Greene Climacteric Scale. Higher Scores indicate higher frequency.
Change Severity of menopause symptoms baseline - interim point | 6 weeks
  Change from baseline severity of menopause symptoms at 6 weeks on a scale from 0 to 3 on the Greene Climacteric Scale. Higher Scores indicate higher severity.
Change Severity of menopause symptoms baseline - endpoint | 12 weeks
  Change from baseline severity of menopause symptoms at 12 weeks on a scale from 0 to 3 on the Greene Climacteric Scale. Higher Scores indicate higher severity.
Change Severity of menopause symptoms interim point - endpoint | 6 weeks
  Change from interim point severity of menopause symptoms at 12 weeks on a scale from 0 to 3 on the Greene Climacteric Scale. Higher Scores indicate higher severity.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Harrison, PhD, Principal Investigator — University of Chester
Locations (1):
- University of Chester, Chester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El Khoudary SR, Aggarwal B, Beckie TM, Hodis HN, Johnson AE, Langer RD, Limacher MC, Manson JE, Stefanick ML, Allison MA; American Heart Association Prevention Science Committee of the Council on Epidemiology and Prevention; and Council on Cardiovascular and Stroke Nursing. Menopause Transition and Cardiovascular Disease Risk: Implications for Timing of Early Prevention: A Scientific Statement From the American Heart Association. Circulation. 2020 Dec 22;142(25):e506-e532. doi: 10.1161/CIR.0000000000000912. Epub 2020 Nov 30. PMID 33251828
- [Result] Gomez-Delgado F, Katsiki N, Lopez-Miranda J, Perez-Martinez P. Dietary habits, lipoprotein metabolism and cardiovascular disease: From individual foods to dietary patterns. Crit Rev Food Sci Nutr. 2021;61(10):1651-1669. doi: 10.1080/10408398.2020.1764487. Epub 2020 Jun 9. PMID 32515660
- [Result] Greene JG. Constructing a standard climacteric scale. Maturitas. 1998 May 20;29(1):25-31. doi: 10.1016/s0378-5122(98)00025-5. PMID 9643514
- [Result] Lobo RA, Gompel A. Management of menopause: a view towards prevention. Lancet Diabetes Endocrinol. 2022 Jun;10(6):457-470. doi: 10.1016/S2213-8587(21)00269-2. Epub 2022 May 5. PMID 35526556
- [Result] Roa-Diaz ZM, Raguindin PF, Bano A, Laine JE, Muka T, Glisic M. Menopause and cardiometabolic diseases: What we (don't) know and why it matters. Maturitas. 2021 Oct;152:48-56. doi: 10.1016/j.maturitas.2021.06.013. Epub 2021 Jul 2. PMID 34674807